CLINICAL TRIAL: NCT02335593
Title: Evaluation of the Effect of Zinc Supplementation on the Health Status of Hemodialysis Patients
Brief Title: Efficacy Study of Zinc Supplementation on Anemia, Oxidative Stress and Inflammation in Hemodialysis Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ain Shams University (Other)
Collaborators: National Institute of Urology and Nephrology (Unknown)
Responsible Party: Principal Investigator, Rasha Roshdy Ibrahim El-kady, Teaching Assistant, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PHCL394
Record Dates: First submitted 2014-12-31; First posted 2015-01-12 (Estimated); Last update posted 2020-01-22 (Actual); Status verified 2020-01

CONDITIONS: End Stage Renal Disease
Keywords: Hemodialysis patients; Zinc; Anemia; Oxidative stress
MeSH Terms: conditions — Kidney Failure, Chronic; Anemia | interventions — Zinc Sulfate; Epoetin Alfa; Solutions; Injections

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Zinc group (Experimental): Zinc Sulphate Hard Gel Capsules 110 mg once daily for three months plus Epoetin alfa 2000-4000 IU solution for injection andIron Hydroxide Saccharate Complex Solution for injection.
  Interventions: Dietary Supplement: Zinc Sulphate; Drug: Epoetin alfa 2000-4000 IU solution for injection; Drug: Iron Hydroxide Saccharate Complex Solution for injection
- Placebo group (Active Comparator): Corn starch filled Hard Gel capsules once daily plus 'Epoetin alfa 2000-4000 IU solution for injection and Iron Hydroxide Saccharate Complex Solution for injection.
  Interventions: Other: Corn Starch filled Hard Gel Capsules; Drug: Epoetin alfa 2000-4000 IU solution for injection; Drug: Iron Hydroxide Saccharate Complex Solution for injection

INTERVENTIONS:
Dietary Supplement: Zinc Sulphate — Zinc Sulphate Hard Gel capsules 110mg
  Arms: Zinc group
Other: Corn Starch filled Hard Gel Capsules — Corn Starch filled Hard Gel Capsules
  Arms: Placebo group
Drug: Epoetin alfa 2000-4000 IU solution for injection — Epoetin alfa 2000-4000 IU solution for injection
Drug: Iron Hydroxide Saccharate Complex Solution for injection — Iron Hydroxide Saccharate Complex Solution for injection

SUMMARY:
The purpose of the study is to evaluate the effect of Zinc supplementation on health status of hemodialysis patients through measurement of the following before and after Zinc administration: Inflammatory markers, Oxidative stress markers and Anemia markers. Also, Evaluation of quality of life of hemodialysis patients before and after Zinc administration using Fatigue severity scale questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* Under regular hemodialysis for at least 6 months.
* Clinically stable condition as outpatients.
* Zinc-deficient patients (plasma Zinc concentrations less than 80 mcg/dl).

Exclusion Criteria:

* Patients taking any antioxidant supplements including vitamin E, Omega-3 fatty acids, green tea preparations or immunosuppressive medications within 2 months prior to enrollment in the study.
* Patients receiving Al hydroxide phosphate binders.
* Hospitalization in the previous month before the onset of the trial, or having active infection.
* Patients with malabsorption diseases (e.g, Crohn's disease), liver diseases, cancers, mental retardation, dementia or psychiatric illness.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2014-12; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Effect on Anemic status (Measurement of Hemoglobin, Hematocrit, serum iron,Total Iron Binding Capacity and serum ferritin) | three months
  at baseline and after 3 monthes.

SECONDARY OUTCOMES:
Effect on Oxidative stress (Measurement of Malondialdehyde, Total antioxidant capacity, Nitric oxide and Superoxide dismutase) | three months
  Measurement of Malondialdehyde, Total antioxidant capacity, Nitric oxide and Superoxide dismutase at baseline and after 3 monthes.
Effect on Inflammatory status. (Measurement of C-Reactive protein and Interleukin-6) | three months
  Measurement of C-Reactive protein and Interleukin-6 at baseline and after 3 monthes.
Effect on Fatigue (Fatigue Sevrity Scale) | three months
  Using Fatigue Sevrity Scale at baseline and after 3 monthes.

CONTACTS AND LOCATIONS:
Overall Officials: Rasha R. El-kady, Bachelor, Principal Investigator — Ain Shams University
Locations (1):
- National Institute of Urology and Nephrology, Cairo, El Matareya, Egypt